CLINICAL TRIAL: NCT01670552
Title: Parallel Study, Double-blind, Randomized, to Compare the Safety of Two Therapies for the Treatment of Osteoarticular Inflammation in Dyspeptic Patients.
Brief Title: Evaluation of Two Therapies for the Treatment of Osteoarticular Inflammation in Dyspeptic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIPEMS1111
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Acute and Chronic Inflammation; Dyspepsia
MeSH Terms: conditions — Dyspepsia | interventions — nimesulide; Pantoprazole; Naproxen; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimesulide + Pantoprazole (Experimental): Nimesulide + Pantoprazole- 1 tablet each 12 hours for 14 days
  Interventions: Drug: Nimesulide + Pantoprazole
- Naproxen + Esomeprazole (Active Comparator): Naproxen + Esomeprazole - 1 tablet each 12 hours for 14 days
  Interventions: Drug: Naproxen + Esomeprazole

INTERVENTIONS:
Drug: Nimesulide + Pantoprazole — 1 tablet each 12 hours for 14 days plus 1 tablet each 12 hours for 14 days of the Naproxen + Esomeprazole placebo.
  Arms: Nimesulide + Pantoprazole
Drug: Naproxen + Esomeprazole — 1 tablet each 12 hours for 14 days plus 1 tablet each 12 hours for 14 days of the Nimesulide + Pantoprazole placebo.
  Other Names: VIMOVO
  Arms: Naproxen + Esomeprazole

SUMMARY:
The purpose of this study is to evaluate the safety of an association with one anti-inflammatory and one gastroprotective agent compared to the one anti-inflammatory and one gastroprotective agent in patients with acute or chronic osteoarticular inflammation.

DETAILED DESCRIPTION:
* Double-blind,randomized, multicenter
* Experiment duration: 14 days
* 03 visits
* Evaluate the safety of an association with one anti-inflammatory and one gastroprotective compared to association with one anti-inflammatory and one gastroprotective agent in patients with acute or chronic osteoarticular inflammation
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

* Adults male or female aged ≥ 18 years old;
* Comply with all the purposes and procedures of the study by signing and dating the Informed Consent.
* Acute or chronic osteo-articular injury in need of of anti-inflammatory for a period of 14 days.

Exclusion Criteria:

* Pregnant women, or women in childbearing age who are not in use effective contraception or intending to become pregnant during the study period
* History of peptic ulcer or gastric surgery;
* Use of Non-steroidal anti-inflammatory (NSAIDs), aspirin, proton pump inhibitor (PPIs), H2 blocker and antacid in the past 7 days;
* Contraindication to the use of NSAIDs or PPIs;
* Renal or hepatic impairment;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2016-02-17 (Actual); Primary Completion 2016-10-28 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Comparison relieve pain in patients with osteoarticular diseases and dyspeptic symptoms, defined as visual analogue scale (VAS) version modified Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). | 14 days

SECONDARY OUTCOMES:
Incidence of adverse events and dyspeptic complaints during the study | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pedro A. Petersen, MD, Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA
Locations (1):
- Allegisa, Campinas, São Paulo, Brazil

REFERENCES:
- [Result] Scheinberg M, Pott Junior H, Macedo EA, Bocchi de Oliveira MF, Ecclissato C, Amazonas RB. Efficacy and safety of a fixed-dose combination of nimesulide/pantoprazole compared to naproxen/esomeprazole for pain relief in patients with osteoarticular diseases and dyspeptic symptoms. Drug Des Devel Ther. 2018 Sep 6;12:2775-2783. doi: 10.2147/DDDT.S172068. eCollection 2018. PMID 30233140